CLINICAL TRIAL: NCT05295030
Title: Effects of Breast Milk Simulated Infant Formula: A 3-month Randomized Controlled Trial
Brief Title: Effects of Breast Milk Simulated Infant Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Huilian Zhu, Professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MN-2022-01
Record Dates: First submitted 2022-03-13; First posted 2022-03-24 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Infant Formula; Breast Milk
Keywords: gut microbiota; temperament; body growth; fecal residual nutrient
MeSH Terms: interventions — Milk, Human

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Breast Milk-Fed Group (Active Comparator): The infants will be breastfed during the study.
  Interventions: Other: Breast milk
- Breast Milk Simulated Formula Group (Experimental): Kieember Infant formula, Ruibuen®: Infants will be fed Kieember infant formula(Phase I) from baseline (1 month old) to 3 month old.
  Interventions: Other: Kieember Infant formula, Ruibuen®
- Traditional Formula Group (Experimental): Yashili Infant formula, Ruibuen®: Infants will be fed Yashili infant formula (Phase I) from baseline (1 month old) to 3 month old.
  Interventions: Other: Yashili Infant formula, Ruibuen®

INTERVENTIONS:
Other: Breast milk — Breast milk: Human breast milk, provided and fed by the corresponding infant's mother
  Arms: Breast Milk-Fed Group
Other: Kieember Infant formula, Ruibuen® — Kieember Infant formula, Ruibuen®: a type of Phase I infant formula for 0-6 month infants, with a trademark of Ruibuen®. The formula is characterized by (1) OPO structured lipid of the third generation; and (2) Breast Milk Simulated complete structured lipid UPU. It was produced by Yashili New Zealand Dairy Co., Limited
  Arms: Breast Milk Simulated Formula Group
Other: Yashili Infant formula, Ruibuen® — Yashili Infant formula, Ruibuen®: a type of Phase I infant formula for 0-6 month infants, with a trademark of Ruibuen®. The formula is characterized by(1) lactoferrin and(2) lutein . It was produced by Yashili International Holdings Ltd.,China
  Arms: Traditional Formula Group

SUMMARY:
Objective：The aim of this trial is to assess effects of Kieember and Yashili infant formula on body growth, behavior development, intestinal comfort, infectious diseases, allergic diseases, the absorption of nutrients and gut microbiota as compared to breast-milk in term infants aged 0-3 months.

Participants：144 healthy term infants aged less than 30 days at entry to study. Study Design: A open-label,parallel, controlled trial.

Arms, Groups, and Intervention: (1) Breast milk-fed group: fed with human breast milk; (2) Breast Milk Simulated Formula Group：fed with breast milk simulated infant formula (Ruibuen®Kieember, Phase I); (3) Traditional Formula Group: fed with traditional infant formula (Ruibuen®Yashili, Phase I).

Intervention Duration: 90 days.

Visits: 1month and 3month old.

Outcome measures: (1)Biochemical detection of feces (total fat, fatty acids, calcium, nitrogen);(2)Stool characteristics (frequency, color, volume, and stool consistency);(3)Anthropometric parameters (body length, body weight, and head circumferences);(4)Temperament and adaptive behavior;(5)Gut microbiota;(6)General health and wellbeing;(7)concomitant medications and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Term infant: Born at 37-42 gestation weeks
* Birth weight: 2500-4000g (appropriate for gestational age)
* The infant is in good health and Apgar after 5 minutes >7
* The mother had unequivocally decided not to breastfeed (for formula fed infants) or to breastfeed (for human milk fed infants)
* age at the enrollment: less than 30 days

Exclusion Criteria:

* The mother is unable to take care of her infant on account of health condition (psychological or physical) or socioeconomic problems
* The infant is born with a congenital malformation or chromosome abnormality with a clinical significance
* The infant suffers from a disease requiring mechanical ventilation or medication in the first week of life (not including applying phototherapy of blue to cure neonatal jaundice)
* The infant whose feeding or normal metabolism is affected by any suspected or unknown metabolic factors or physical limitations
* The infant has been breastfed for more than 2 weeks (for formula fed infants)
* Twins or multiple births

Ages: 0 Days to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 179 (Actual)
Dates: Start 2022-04-10 (Actual); Primary Completion 2023-12-25 (Actual); Study Completion 2023-12-25 (Actual)

PRIMARY OUTCOMES:
Average Change Rate of Gut Microbiota Pattern Score from 1month to 3 month | 1,3 months
  Slope of change at 1 and 3 month in gut microbiota pattern score from 16S RNA sequencing.
Average Change Rate of Fecal Residual Fatty Acid from 1month to 3 month | 1,3 months
  Slope of change at 1 and 3 month in Fecal Residual Fatty Acid.
Average Change Rate of Fecal Residual Nitrogen from 1month to 3 month | 1,3 months
  Slope of change at 1 and 3 month in Fecal Residual Nitrogen.
Average Change Rate of Fecal Residual Calcium from 1month to 3 month | 1,3 months
  Slope of change at 1 and 3 month in fecal residual calcium.
Average Change Rate of body length from 1month to 3 month | 1,3 months
  Slope of change at 1 and 3 month in body length.
Average Change Rate of body weight from 1month to 3 month | 1,3 months
  Slope of change at 1 and 3 month in body weigh.
Average Change Rate of head circumferences from 1month to 3 month | 1,3 months
  Slope of change at 1 and 3 month in head circumferences.

SECONDARY OUTCOMES:
Average Change Rate of Stool Characteristic Index from 1month to 3 month | 1,3 months
  Slope of change at 1 and 3 month in Stool Characteristic Index: calculated by using stool color (using sample pictures), stool shape (using sample pictures), and frequency.
Average Change Rate of an Index of General health and wellbeing from 1month to 3 month | 1,3 months
  Slope of change at 1 and 3 month in Index of General health and wellbeing, calculated from diseases (cold, diarrhea,infectious diseases), doctor visits, concomitant medications,etc.
Average Change Rate of Temperament Score from 1month to 3 month | 1,3 months
  Slope of change at 1 and 3 month in Temperament Score assessed by the Early Infant Temperament Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China